CLINICAL TRIAL: NCT03179176
Title: Evaluation of the Interest of Ultra-high Frequency Doppler Ultrasound (UFDU) in the Surgical Management of Patients Operated in an Awake Condition for a Cerebral Tumor
Acronym: EUHF_PRC
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Centre Hospitalier Universitaire de Nice (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: 17-PP-01
Record Dates: First submitted 2017-05-29; First posted 2017-06-07 (Actual); Last update posted 2024-02-06 (Actual); Status verified 2024-02

CONDITIONS: Cerebral Tumor

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- HFUD utilisation (Experimental)
  Interventions: Other: High Frequence Ultrasound Doppler (HFUD) utilisation

INTERVENTIONS:
Other: High Frequence Ultrasound Doppler (HFUD) utilisation — Utilisation of HFUD will be done during on patients during an operation in waking condition. This procedure extends the usual procedure from 15 to 20 minutes.

SUMMARY:
In brain tumor surgery we are confronted mainly with two types of difficulties: (i) the identification of the tumor and its limitations in relation to the healthy brain; (ii) the identification of functional cerebral regions, ie implicated in neurological function (motor skills, sensitivity, language, vision, cognition, etc.). The reference method currently used to improve the quality of resection of brain tumors while minimizing neurological risk for patients is so called "wakeful" surgery with direct electrical stimulation (DES) of the brain. The investigators routinely use ultrasound to localize the tumor within the brain, but to date there is no pre- or intra-operative imaging tool to reliably identify tumors and functional brain regions. There is therefore a need for innovative imaging in this field.

For this reason, the investigators propose to evaluate the interest of a new High Frequence Ultrasound Doppler (HFUD) (VEVO ®, Visualsonics, Toronto, Canada) in the surgical management of patients operated in an awake condition for a brain tumor. The ultra high frequency allows to reach a spatial resolution of 30 μm, 5 to 10 times better than MRI and conventional ultrasound. The Doppler mode allows the detection of microvascular flows of speeds less than 1 mm / second. The safety of this device is demonstrated and validated by CE marking (December 2015).

ELIGIBILITY:
Inclusion Criteria:

* operated patient of a cerebral tumor in an awake condition
* age> 18 years
* neurological condition allowing the realization of the tests in the operating room

Exclusion Criteria:

* not indicated for "awake" surgery
* refusal of participation of the patient
* pregnant or nursing women

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 4 (Actual)
Dates: Start 2017-04-25 (Actual); Primary Completion 2018-04-25 (Actual); Study Completion 2018-04-25 (Actual)

PRIMARY OUTCOMES:
Diameter of the sulcus blood vessels | before resection of the tumor

CONTACTS AND LOCATIONS:
Overall Officials: Fabien ALMAIRAC, MD, Study Director — Centre Hospitalier Universitaire de Nice
Locations (1):
- CHU de Nice, Nice, France

REFERENCES:
- [Derived] Almairac F, Fontaine D, Demarcy T, Delingette H, Beuil S, Raffaelli C. Motor cortex neurovascular coupling: inputs from ultra-high-frequency ultrasound imaging in humans. J Neurosurg. 2018 Nov 9;131(5):1632-1638. doi: 10.3171/2018.5.JNS18754. Print 2019 Nov 1. PMID 30497179